CLINICAL TRIAL: NCT01180790
Title: A Phase IIa, Randomized, Double-blind (Participant and Investigator Blind, Sponsor Open), Placebo-controlled Trial to Evaluate the Safety, Tolerability, and Antiviral Activity of Oral ACH-0141625 in Combination With Pegylated Interferon Alpha-2a and Ribavirin in Two Segments, After 28 Days of Dosing and, Subsequently, After 12 Weeks of Dosing in Participants With Chronic Hepatitis C Virus Genotype 1
Brief Title: Safety, Tolerability, and Antiviral Activity of ACH-0141625 or Placebo in Combination With Peginterferon and Ribavirin in Hepatitis C Virus (HCV) Positive Participants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: Achillion, a wholly owned subsidiary of Alexion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACH625-003; 2010-022092-65 (EudraCT Number)
Record Dates: First submitted 2010-08-11; First posted 2010-08-12 (Estimated); Results first posted 2014-09-10 (Estimated); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Hepatitis C
Keywords: HCV; Hepatitis C Genotype 1
MeSH Terms: conditions — Hepatitis C | interventions — peginterferon alfa-2a; peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (7):
- Segment 1: 200 milligrams (mg) ACH-0141625 (Experimental): 200 mg ACH-0141625 for 28 days plus pegylated interferon (Peg-IFN) alpha-2a and ribavirin (RBV) for 48 weeks
  Interventions: Drug: ACH-0141625 (Sovaprevir); Drug: Pegylated Interferon alpha-2a; Drug: Ribavirin
- Segment 1: 400 mg ACH-0141625 (Experimental): 400 mg ACH-0141625 for 28 days plus Peg-IFN alpha-2a plus RBV for 48 weeks
  Interventions: Drug: ACH-0141625 (Sovaprevir); Drug: Pegylated Interferon alpha-2a; Drug: Ribavirin
- Segment 1: 800 mg ACH-0141625 (Experimental): 800 mg ACH-0141625 for 28 days plus Peg-IFN alpha-2a plus RBV for 48 weeks
  Interventions: Drug: ACH-0141625 (Sovaprevir); Drug: Pegylated Interferon alpha-2a; Drug: Ribavirin
- Segment 1: Placebo (Placebo Comparator): Placebo for 28 days plus Peg-IFN alpha-2a plus RBV for 48 weeks
  Interventions: Drug: Placebo; Drug: Pegylated Interferon alpha-2a; Drug: Ribavirin
- Segment 2: 200 mg ACH-0141625 (Experimental): 200 mg ACH-0141625 for 12 weeks plus Peg-IFN and RBV for up to a total of 24 or 48 weeks
  Interventions: Drug: ACH-0141625 (Sovaprevir); Drug: Pegylated Interferon alpha-2a; Drug: Ribavirin
- Segment 2 : 400 mg ACH-0141625 (Experimental): 400 mg ACH-0141625 for 12 weeks plus Peg-IFN and RBV for up to a total of 24 or 48 weeks
  Interventions: Drug: ACH-0141625 (Sovaprevir); Drug: Pegylated Interferon alpha-2a; Drug: Ribavirin
- Segment 2 : 800 mg ACH-0141625 (Experimental): 800 mg ACH-0141625 for 12 weeks plus Peg-IFN and RBV for up to a total of 24 or 48 weeks
  Interventions: Drug: ACH-0141625 (Sovaprevir); Drug: Pegylated Interferon alpha-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: ACH-0141625 (Sovaprevir) — 200 mg oral capsule once daily
  Arms: Segment 1: 200 milligrams (mg) ACH-0141625; Segment 2: 200 mg ACH-0141625
Drug: ACH-0141625 (Sovaprevir) — 400 mg oral capsule once daily
  Arms: Segment 1: 400 mg ACH-0141625; Segment 2 : 400 mg ACH-0141625
Drug: ACH-0141625 (Sovaprevir) — 800 mg oral capsule once daily
  Arms: Segment 1: 800 mg ACH-0141625; Segment 2 : 800 mg ACH-0141625
Drug: Placebo — Powder in capsule once daily
  Arms: Segment 1: Placebo
Drug: Pegylated Interferon alpha-2a — 180 micrograms (ug) once a week by subcutaneous injection
  Other Names: Peg-INF
Drug: Ribavirin — 400 mg or 600 mg (morning [AM]) and 600 mg (evening [PM]) capsules taken orally twice daily
  Other Names: Ribasphere; Copegus

SUMMARY:
Evaluate safety, tolerability, and antiviral response of ACH-0141625 compared to standard of care in hepatitis C virus (HCV)-positive participants.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, aged 18 years and older
* Chronic hepatitis C genotype 1 (as specified in the protocol)
* Treatment naive
* Females who are post-menopausal and amenorrheic must have a follicle-stimulating hormone (FSH) at screening. Females of childbearing potential must have a negative pregnancy test at screening and baseline. Females must use a non-hormonal method of contraception and must agree not to get pregnant during the study and for 6 months following the discontinuation of standard of care (SOC).
* Fertile males must agree to use a condom and his female partner must agree to use 1 or more methods of contraception. Males must not donate sperm during the study and 3 months following the last exposure to RBV.

Exclusion Criteria:

* Body mass index (BMI) >36 kilograms (kg)/square meter (m^2)
* Pregnant or nursing females or females of childbearing potential not willing to comply with contraceptive measures per protocol. Men whose female partners are pregnant or contemplating pregnancy. - Coinfection with hepatitis B virus (HBV) and/or human immunodeficiency virus (HIV)
* Other significant diseases including liver disease
* History of drug or alcohol dependence or addiction within the past 6 months
* History of participation in a clinical trial with a protease inhibitor or previous treatment with a protease inhibitor, where at least 1 dose of the protease inhibitor was consumed.
* Use of herbal or homeopathic products, illicit drugs, cytochrome P450 (CYP) 3A4/5 substrates, inducers or inhibitors, hormonal methods of contraception, corticosteroids, immunosuppressive, or cytotoxic agents within 28 days of the first dose of study drug.
* Have a clinically significant laboratory abnormality at screening (as specified in the protocol).
* Segment 1: Participants with any history of decompensated liver disease defined as cirrhotic participants with a Child-Pugh score of > or = to 7. Segment 2: Participants who have had a liver biopsy that shows bridging fibrosis or cirrhosis.
* Nonalcoholic steatohepatitis if ballooning degeneration or Mallory bodies are present on liver biopsy.
* Participants who prematurely discontinued, interrupted, or dose reduced prior Peg-IFN and RBV therapy due to noncompliance or safety issues.
* Encephalopathy or altered mental status of any etiology.
* History of moderate, severe, or uncontrolled psychiatric disease (as specified in the protocol).
* History of malignancy of any organ system treated or untreated within the past 5 years.
* Use of colony stimulating factor agents within 90 days prior to baseline.
* History of seizure disorder.
* History of known coagulopathy including hemophilia.
* Clinically of significant findings on fundoscopic or retinal examination at screening
* History of immunologically mediate disease.
* History of clinical evidence of chronic cardiac disease (as specified in the protocol)
* Received concomitant systemic antibiotic, antifungals, or antivirals for the treatment of active infection within 14 days prior to the first dose of the study drug (as specified in the protocol)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2010-09; Primary Completion 2012-03 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (14):
  - Clinical Trial Site, Los Angeles, California
  - Clinical Trial Site, San Francisco, California
  - Clinical Trial Site, Bradenton, Florida
  - Clinical Trial Site, Orlando, Florida
  - Clinical Trial Site, Chicago, Illinois
  - Clinical Trial Site, Overland Park, Kansas
  - Clinical Trial Site, St Louis, Missouri
  - Clinical Trial Site, Las Vegas, Nevada
  - Clinical Trial Site, New York, New York
  - Clinical Trial Site, Philadelphia, Pennsylvania
  - Clinical Trial Site, Arlington, Texas
  - Clinical Trial Site, San Antonio, Texas
  - Clinical Trial Site, Newport News, Virginia
  - Clinical Trial Site, Norfolk, Virginia
- Belgium (3):
  - Clinical Trial Site, Edegem, Antwerp
  - Clinical Trial Site, Haine-Saint-Paul, Hainaut
  - Clinical Trial Site, Ghent, Oost-Vlaanderen

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 15 sites in the United States and 3 sites in Belgium between 30 September 2010 and 03 January 2012.
Pre-assignment Details: Participants were screened within 4 weeks (Day -28 to Day -1) before administration of the study drug. Participants who meet all eligibility criteria were instructed to arrive at the study center on Baseline day for randomization to treatment assignment.
Groups:
- Segment 1: 200 Milligrams (mg) ACH-0141625 for 28 Days: ACH-0141625: 200 mg oral capsule once daily
  Pegylated Interferon (Peg-IFN) alpha-2a: 180 micrograms (ug) once a week by subcutaneous injection for 48 weeks
  Ribavirin (RBV): 400 mg or 600 mg (morning [AM]) and 600 mg (evening [PM]) capsules taken orally twice daily for 48 weeks
- Segment 1: 400 mg ACH-0141625 for 28 Days: ACH-0141625: 400 mg oral capsule once daily
  Peg-IFN alpha-2a: 180 ug once a week by subcutaneous injection for 48 weeks
  RBV: 400 mg or 600 mg (AM) and 600 mg (PM) capsules taken orally twice daily for 48 weeks
- Segment 1: 800 mg ACH-0141625 for 28 Days: ACH-0141625: 800 mg oral capsule once daily
  Peg-IFN alpha-2a: 180 ug once a week by subcutaneous injection for 48 weeks
  RBV: 400 mg or 600 mg (AM) and 600 mg (PM) capsules taken orally twice daily for 48 weeks
- Segment 1: Placebo for 28 Days: Placebo: Powder in capsule once daily
  Peg-IFN alpha-2a: 180 ug once a week by subcutaneous injection for 48 weeks
  RBV: 400 mg or 600 mg (AM) and 600 mg (PM) capsules taken orally twice daily for 48 weeks
- Segment 2: 200 mg ACH-0141625 for 12 Weeks: ACH-0141625: 200 mg oral capsule once daily
  Peg-IFN alpha-2a: 180 ug once a week by subcutaneous injection for up to 24 or 48 weeks
  RBV: 400 mg or 600 mg (AM) and 600 mg (PM) capsules taken orally twice daily for up to 24 or 48 weeks
- Segment 2: 400 mg ACH-0141625 for 12 Weeks: ACH-0141625: 400 mg oral capsule once daily
  Peg-IFN alpha-2a: 180 ug once a week by subcutaneous injection for up to 24 or 48 weeks
  RBV: 400 mg or 600 mg (AM) and 600 mg (PM) capsules taken orally twice daily for up to 24 or 48 weeks
- Segment 2: 800 mg ACH-0141625 for 12 Weeks: ACH-0141625: 800 mg oral capsule once daily
  Peg-IFN alpha-2a: 180 ug once a week by subcutaneous injection for up to 24 or 48 weeks
  RBV: 400 mg or 600 mg (AM) and 600 mg (PM) capsules taken orally twice daily for up to 24 or 48 weeks
Period: Overall Study
Arm/Group | Segment 1: 200 Milligrams (mg) ACH-0141625 for 28 Days | Segment 1: 400 mg ACH-0141625 for 28 Days | Segment 1: 800 mg ACH-0141625 for 28 Days | Segment 1: Placebo for 28 Days | Segment 2: 200 mg ACH-0141625 for 12 Weeks | Segment 2: 400 mg ACH-0141625 for 12 Weeks | Segment 2: 800 mg ACH-0141625 for 12 Weeks
Started | 16 | 16 | 17 | 15 | 19 | 20 | 19
Completed | 7 | 11 | 4 | 6 | 14 | 13 | 18
Not Completed | 9 | 5 | 13 | 9 | 5 | 7 | 1
Not completed — Adverse Event | 1 | 1 | 2 | 0 | 1 | 3 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 5 | 0 | 2 | 1 | 0
Not completed — Lost to Follow-up | 3 | 1 | 0 | 2 | 1 | 0 | 1
Not completed — Physician Decision | 1 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 2 | 5 | 6 | 1 | 3 | 0
Not completed — compliance | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Severe coronary atherosclerosis (death) | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population, which was defined as all participants randomized and treated with at least 1 dose of ACH 0141625 or Placebo. Participants were analyzed according to the randomized treatment.
Groups:
- Segment 1: 200 mg ACH-0141625: 200 mg ACH-0141625 for 28 days plus Peg-IFN alpha-2a and RBV for 48 weeks
  ACH-0141625: 200 mg oral capsule once daily for 28 days or for 12 weeks
  Peg-IFN alpha-2a: 180 ug once a week by subcutaneous injection for 48 weeks
  RBV: 400 mg or 600 mg (AM) and 600 mg (PM) capsules taken orally twice daily for 48 weeks
- Segment 1: 400 mg ACH-0141625: 400 mg ACH-0141625 for 28 days plus Peg-IFN alpha-2a plus RBV for 48 weeks
  ACH-0141625: 400 mg oral capsule once daily for 28 days or for 12 weeks
  Peg-IFN alpha-2a: 180 ug once a week by subcutaneous injection for 48 weeks
  RBV: 400 mg or 600 mg (AM) and 600 mg (PM) capsules taken orally twice daily for 48 weeks
- Segment 1: 800 mg ACH-0141625: 800 mg ACH-0141625 for 28 days plus Peg-IFN alpha-2a plus RBV for 48 weeks
  ACH-0141625: 800 mg oral capsule once daily for 28 days or for 12 weeks
  Peg-IFN alpha-2a: 180 ug once a week by subcutaneous injection for 48 weeks
  RBV: 400 mg or 600 mg (AM) and 600 mg (PM) capsules taken orally twice daily for 48 weeks
- Segment 1: Placebo: Placebo for 28 days plus Peg-IFN alpha-2a plus RBV for 48 weeks
  Placebo: Powder in capsule once daily for 28 days
  Peg-IFN alpha-2a: 180 ug once a week by subcutaneous injection for 48 weeks
  RBV: 400 mg or 600 mg (AM) and 600 mg (PM) capsules taken orally twice daily for 48 weeks
- Segment 2: 200 mg ACH-0141625: 200 mg ACH-0141625 for 12 weeks plus Peg-IFN and RBV for up to a total of 48 weeks
  ACH-0141625: 200 mg oral capsule once daily for 28 days or for 12 weeks
  Peg-IFN alpha-2a: 180 ug once a week by subcutaneous injection for 48 weeks
  RBV: 400 mg or 600 mg (AM) and 600 mg (PM) capsules taken orally twice daily for 48 weeks
- Segment 2: 400 mg ACH-0141625: 400 mg ACH-0141625 for 12 weeks plus Peg-IFN and RBV for up to a total of 48 weeks
  ACH-0141625: 400 mg oral capsule once daily for 28 days or for 12 weeks
  Peg-IFN alpha-2a: 180 ug once a week by subcutaneous injection for 48 weeks
  RBV: 400 mg or 600 mg (AM) and 600 mg (PM) capsules taken orally twice daily for 48 weeks
- Segment 2: 800 mg ACH-0141625: 800 mg ACH-0141625 for 12 weeks plus Peg-IFN and RBV for up to a total of 48 weeks
  ACH-0141625: 800 mg oral capsule once daily for 28 days or for 12 weeks
  Peg-IFN alpha-2a: 180 ug once a week by subcutaneous injection for 48 weeks
  RBV: 400 mg or 600 mg (AM) and 600 mg (PM) capsules taken orally twice daily for 48 weeks
- Total: Total of all reporting groups
Arm/Group | Segment 1: 200 mg ACH-0141625 | Segment 1: 400 mg ACH-0141625 | Segment 1: 800 mg ACH-0141625 | Segment 1: Placebo | Segment 2: 200 mg ACH-0141625 | Segment 2: 400 mg ACH-0141625 | Segment 2: 800 mg ACH-0141625 | Total
Number analyzed (Participants) | 16 | 16 | 17 | 15 | 19 | 20 | 19 | 122
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 16 | 16 | 15 | 19 | 19 | 19 | 119
  >=65 years | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (7) | 51 (9) | 52 (13) | 47 (9) | 45 (11) | 48 (12) | 42 (12) | 48 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 4 | 4 | 7 | 5 | 9 | 38
  Male | 13 | 10 | 13 | 11 | 12 | 15 | 10 | 84

OUTCOME MEASURES:

1. Primary Outcome: Segment 1: Safety
Description: Segment 1: Percentage of participants with the following: adverse events, abnormal laboratory safety tests, dose reductions, interruptions, and discontinuations. Criteria for abnormal laboratory safety tests: treatment-emergent worsening Division of AIDS (Acquired Immunodeficiency Syndrome) (DAIDs) graded laboratory tests. A summary of serious and all other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: 4 weeks
Population: The safety population, which was defined as all participants randomized and treated with at least one dose of ACH-0141625 or Placebo. Participants were analyzed according to the randomized treatment.
Measure: Number; unit: percentage of participants
Groups:
- Segment 1: Placebo: Placebo for 28 days plus Peg-IFN alpha-2a plus ribavirin for 48 weeks
  Placebo: Powder in capsule once daily
  Pegylated Interferon alpha-2a: 180 ug once a week by subcutaneous injection
  ribavirin: 400 mg or 600 mg (am) and 600 mg (pm) capsules taken orally twice daily
- Segment 1: 200 mg ACH-0141625: 200 mg ACH-0141625 for 28 days plus Peg-IFN alpha-2a and ribavirin for 48 weeks
  ACH-0141625: 200 mg oral capsule once daily
  Pegylated Interferon alpha-2a: 180 ug once a week by subcutaneous injection for
  ribavirin: 400 mg or 600 mg (am) and 600 mg (pm) capsules taken orally twice daily
- Segment 1: 400 mg ACH-0141625: 400 mg ACH-0141625 for 28 days plus Peg-IFN alpha-2a plus ribavirin for 48 weeks
  ACH-0141625: 400 mg oral capsule once daily
  Pegylated Interferon alpha-2a: 180 ug once a week by subcutaneous injection
  ribavirin: 400 mg or 600 mg (am) and 600 mg (pm) capsules taken orally twice daily
- Segment 1: 800 mg ACH-0141625: 800 mg ACH-0141625 for 28 days plus Peg-IFN alpha-2a plus ribavirin for 48 weeks
  ACH-0141625: 800 mg oral capsule once daily
  Pegylated Interferon alpha-2a: 180 ug once a week by subcutaneous injection
  ribavirin: 400 mg or 600 mg (am) and 600 mg (pm) capsules taken orally twice daily
Arm/Group | Segment 1: Placebo | Segment 1: 200 mg ACH-0141625 | Segment 1: 400 mg ACH-0141625 | Segment 1: 800 mg ACH-0141625
Number analyzed (Participants) | 15 | 16 | 16 | 17
percentage of participants
  Adverse Events (%) | 93.3 | 100.0 | 93.8 | 100.0
  Abnormal Laboratories (%) | 100.0 | 100.0 | 100.0 | 94.0
  Dose Reductions (%) | 0 | 0 | 0 | 0
  Dose Interruptions (%) | 0 | 0 | 0 | 0
  Dose Discontinuations (%) | 0 | 6.0 | 0 | 6.0

2. Primary Outcome: Segment 1: Rapid Viral Response At Week 4 (RVR4)
Description: The primary efficacy endpoint for Segment 1 of the study was the percentage of participants in each treatment group achieving RVR4 (hepatitis C virus [HCV] ribonucleic acid (RNA) less than or equal to the limit of quantitation [LOQ] at the Week 4 visit).
Time Frame: 4 weeks
Population: Efficacy analysis was performed on the virology population (a subset of the ITT population) and included all participants who had a baseline HCV RNA result and at least 1 post-baseline HCV RNA result.
Measure: Number; unit: percentage of participants
Groups:
- Segment 1: Placebo: Placebo for 28 days plus Peg-IFN alpha-2a plus RBV for 48 weeks
  Placebo: Powder in capsule once daily
  Peg-IFN alpha-2a: 180 ug once a week by subcutaneous injection
  RBV: 400 mg or 600 mg (AM) and 600 mg (PM) capsules taken orally twice daily
- Segment 1: 200 mg ACH-0141625: 200 mg ACH-0141625 for 28 days plus Peg-IFN alpha-2a and RBV for 48 weeks
  ACH-0141625: 200 mg oral capsule once daily
  Peg-IFN alpha-2a: 180 ug once a week by subcutaneous injection
  RBV: 400 mg or 600 mg (AM) and 600 mg (PM) capsules taken orally twice daily
- Segment 1: 400 mg ACH-0141625: 400 mg ACH-0141625 for 28 days plus Peg-IFN alpha-2a plus RBV for 48 weeks
  ACH-0141625: 400 mg oral capsule once daily
  Peg-IFN alpha-2a: 180 ug once a week by subcutaneous injection
  RBV: 400 mg or 600 mg (AM) and 600 mg (PM) capsules taken orally twice daily
- Segment 1: 800 mg ACH-0141625: 800 mg ACH-0141625 for 28 days plus Peg-IFN alpha-2a plus RBV for 48 weeks
  ACH-0141625: 800 mg oral capsule once daily
  Peg-IFN alpha-2a: 180 ug once a week by subcutaneous injection
  RBV: 400 mg or 600 mg (AM) and 600 mg (PM) capsules taken orally twice daily
Arm/Group | Segment 1: Placebo | Segment 1: 200 mg ACH-0141625 | Segment 1: 400 mg ACH-0141625 | Segment 1: 800 mg ACH-0141625
Number analyzed (Participants) | 15 | 16 | 16 | 17
percentage of participants
  Rapid Virologic Response (%) | 20.0 | 75.0 | 75.0 | 76.5
  No Rapid Virologic Response (%) | 80.0 | 25.0 | 25.0 | 23.5
Statistical Analysis 1: Comparison: Segment 1: Placebo vs Segment 1: 200 mg ACH-0141625 vs Segment 1: 400 mg ACH-0141625 vs Segment 1: 800 mg ACH-0141625; The null hypothesis is no difference between proportions of participants in each treatment group achieving RVR4 at Week 4 of the study, while the alternative hypothesis is that the proportion of participants achieving RVR4 at Week 4 increases with increasing doses of ACH-0141625; Test type: Superiority or Other; p = 0.003, exact Cochran-Armitage test — To control for multiplicity, the proportion in each treatment group achieving RVR4 is analyzed using a Cochran-Armitage test for trend among the ordered groups: placebo (considered zero dose), 200 mg, 400 mg, and 800 mg ACH-0141625; Only if overall test for trend is significant are pairwise comparisons evaluated using p-values for the difference in proportions (placebo - active)
Statistical Analysis 2: Comparison: Segment 1: Placebo vs Segment 1: 200 mg ACH-0141625; To control for multiplicity, the proportion in each treatment group achieving RVR4 is analyzed using a Cochran-Armitage test for trend among the ordered groups: placebo (considered zero dose), 200 mg ACH-0141625, 400 mg ACH-0141625, and 800 mg ACH-0141625. Only if overall test for trend is significant are pairwise comparisons evaluated using p-values for the difference in proportions (placebo - active); Test type: Superiority or Other; p = 0.004, Fisher Exact
Statistical Analysis 3: Comparison: Segment 1: Placebo vs Segment 1: 400 mg ACH-0141625; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.004, Fisher Exact
Statistical Analysis 4: Comparison: Segment 1: Placebo vs Segment 1: 800 mg ACH-0141625; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.004, Fisher Exact

3. Primary Outcome: Segment 2: Safety
Description: Segment 2: Percentage of participants with the following: adverse events, abnormal laboratory safety tests and dose reductions, interruptions and discontinuations. Criteria for abnormal laboratory safety tests: treatment-emergent worsening DAIDs graded laboratory tests. A summary of serious and all other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: 12 weeks
Population: The safety population, which was defined as all participants randomized and treated with at least 1 dose of ACH-0141625. Participants were analyzed according to the randomized treatment.
Measure: Number; unit: percentage of participants
Groups:
- Segment 2: 200 mg ACH-0141625: 200 mg ACH-0141625 for 12 weeks plus Peg-IFN alpha-2a and RBV for up to a total of 24 or 48 weeks
  ACH-0141625: 200 mg oral capsule once daily
  Peg-IFN alpha-2a: 180 ug once a week by subcutaneous injection
  RBV: 400 mg or 600 mg (AM) and 600 mg (PM) capsules taken orally twice daily
- Segment 2: 400 mg ACH-0141625: 400 mg ACH-0141625 for 12 weeks plus Peg-IFN alpha-2a plus RBV for up to 24 or 48 weeks
  ACH-0141625: 400 mg oral capsule once daily
  Peg-IFN alpha-2a: 180 ug once a week by subcutaneous injection
  RBV: 400 mg or 600 mg (AM) and 600 mg (PM) capsules taken orally twice daily
- Segment 2: 800 mg ACH-0141625: 800 mg ACH-0141625 for 12 weeks plus Peg-IFN alpha-2a plus RBV for up to 24 or 48 weeks
  ACH-0141625: 800 mg oral capsule once daily
  Peg-IFN alpha-2a: 180 ug once a week by subcutaneous injection
  RBV: 400 mg or 600 mg (AM) and 600 mg (PM) capsules taken orally twice daily
Arm/Group | Segment 2: 200 mg ACH-0141625 | Segment 2: 400 mg ACH-0141625 | Segment 2: 800 mg ACH-0141625
Number analyzed (Participants) | 19 | 20 | 19
percentage of participants
  Adverse Events (%) | 94.7 | 85.0 | 100.0
  Abnormal Laboratories (%) | 100.0 | 95.0 | 100.0
  Dose Reductions (%) | 0 | 0 | 0
  Dose Interruptions (%) | 0 | 0 | 0
  Dose Discontinuations (%) | 6.0 | 20.0 | 0

4. Primary Outcome: Segment 2: Complete Early Virologic Response (cEVR)
Description: The primary efficacy endpoint for Segment 2 of the study was the percentage of participants achieving cEVR, defined as undetectable HCV RNA at Week 12.
Time Frame: Week 12
Population: Per protocol virology population (a subset of the virology population) and included all randomized participants who completed 12 weeks of ACH-0141625 dosing.
Measure: Number; unit: percentage of participants
Groups:
- Segment 2: 200 mg ACH-0141625: 200 mg ACH-0141625 for 12 weeks plus Peg-IFN and RBV for up to a total of 24 or 48 weeks
  ACH-0141625: 200 mg oral capsule once daily
  Peg-IFN alpha-2a: 180 ug once a week by subcutaneous injection
  RBV: 400 mg or 600 mg (AM) and 600 mg (PM) capsules taken orally twice daily
- Segment 2: 400 mg ACH-0141625: 400 mg ACH-0141625 for 12 weeks plus Peg-IFN and RBV for up to a total of 24 or 48 weeks
  ACH-0141625: 400 mg oral capsule once daily
  Peg-IFN alpha-2a: 180 ug once a week by subcutaneous injection
  RBV: 400 mg or 600 mg (AM) and 600 mg (PM) capsules taken orally twice daily
- Segment 2: 800 mg ACH-0141625: 800 mg ACH-0141625 for 12 weeks plus Peg-IFN and RBV for up to a total of 24 or 48 weeks
  ACH-0141625: 800 mg oral capsule once daily for 28 days
  Peg-IFN alpha-2a: 180 ug once a week by subcutaneous injection
  RBV: 400 mg or 600 mg (AM) and 600 mg (PM) capsules taken orally twice daily
Arm/Group | Segment 2: 200 mg ACH-0141625 | Segment 2: 400 mg ACH-0141625 | Segment 2: 800 mg ACH-0141625
Number analyzed (Participants) | 18 | 16 | 19
percentage of participants | 100.0 | 94.0 | 100.00
Statistical Analysis 1: Comparison: Segment 2: 200 mg ACH-0141625 vs Segment 2: 400 mg ACH-0141625 vs Segment 2: 800 mg ACH-0141625; The null hypothesis is no difference between proportions of participants in each treatment group achieving cEVR at Week 12 of the study, while the alternative hypothesis is that the proportion of participants achieving cEVR at Week 12 increases with increasing doses of ACH-0141625; Test type: Superiority or Other; p = 0.34, Exact Cochran-Armitage test — To control for multiplicity, the proportion of participants in each treatment group achieving cEVR is analyzed using a Cochran-Armitage test for trend among the ordered treatment groups: 200 mg ACH-0141625, 400 mg ACH-0141625, and 800 mg ACH-0141625; [statistical method as in outcome 2, analysis 1]

5. Secondary Outcome: Segment 1: cEVR
Description: For Segment 1, the percentage of participants in the virology population who achieved cEVR, defined as undetectable HCV RNA at Week 12.
Time Frame: 12 weeks
Population: Analysis for Segment 1 was performed on the virology population (the same as the ITT population) and included all participants who had a baseline HCV RNA result and at least 1 post-baseline HCV RNA result.
Measure: Number; unit: percentage of participants
Arm/Group | Segment 1: 200 mg ACH-0141625 | Segment 1: 400 mg ACH-0141625 | Segment 1: 800 mg ACH-0141625 | Segment 1: Placebo
Number analyzed (Participants) | 16 | 16 | 17 | 15
percentage of participants | 62.5 | 75.0 | 70.6 | 33.3

6. Secondary Outcome: Segment 2: RVR4
Description: For Segment 2, the percentage of participants in the virology population who achieved RVR4, defined as HCV RNA less than or equal to the LOQ at the Week 4 visit.
Time Frame: 4 weeks
Population: Per protocol virology population (a subset of the virology population) and included all randomized participants who completed 4 weeks of ACH-0141625 dosing.
Measure: Number; unit: percentage of participants
Groups:
- Segment 2: 200 mg ACH-0141625: 200 mg ACH-0141625 for 12 weeks plus Peg-IFN alpha-2a and RBV for 48 weeks
  ACH-0141625: 200 mg oral capsule once daily for 28 days or for 12 weeks
  Peg-IFN alpha-2a: 180 ug once a week by subcutaneous injection for 48 weeks
  RBV: 400 mg or 600 mg (AM) and 600 mg (PM) capsules taken orally twice daily for 48 weeks
- Segment 2: 400 mg ACH-0141625: 400 mg ACH-0141625 for 12 weeks plus Peg-IFN alpha-2a plus RBV for 48 weeks
  ACH-0141625: 400 mg oral capsule once daily for 28 days or for 12 weeks
  Peg-IFN alpha-2a: 180 ug once a week by subcutaneous injection for 48 weeks
  RBV: 400 mg or 600 mg (AM) and 600 mg (PM) capsules taken orally twice daily for 48 weeks
- Segment 2: 800 mg ACH-0141625: 800 mg ACH-0141625 for 12 weeks plus Peg-IFN alpha-2a plus RBV for 48 weeks
  ACH-0141625: 800 mg oral capsule once daily for 28 days or for 12 weeks
  Peg-IFN alpha-2a: 180 ug once a week by subcutaneous injection for 48 weeks
  RBV: 400 mg or 600 mg (AM) and 600 mg (PM) capsules taken orally twice daily for 48 weeks
Arm/Group | Segment 2: 200 mg ACH-0141625 | Segment 2: 400 mg ACH-0141625 | Segment 2: 800 mg ACH-0141625
Number analyzed (Participants) | 19 | 18 | 19
percentage of participants | 78.9 | 88.8 | 89.5

7. Secondary Outcome: Segment 1 And Segment 2: End Of Treatment Response
Description: The percentage of virology population participants who were reported as undetectable HCV RNA at the completion of treatment.
Time Frame: Week 48 (Segment 1); Week 24 (Segment 2)
Population: Segment 2 analyzed the per protocol population (PPP), which includes all randomized participants who completed 12 weeks of ACH-0141625 dosing and an additional 12 weeks of Peg/RBV dosing.
Measure: Number; unit: percentage of participants
Groups:
- Segment 2: 800 mg ACH-0141625: 800 mg ACH-0141625 for 12 weeks plus Peg-IFN and RBV for up to a total of 24 or 48 weeks
  ACH-0141625: 800 mg oral capsule once daily
  Peg-IFN alpha-2a: 180 ug once a week by subcutaneous injection
  RBV: 400 mg or 600 mg (AM) and 600 mg (PM) capsules taken orally twice daily
Arm/Group | Segment 1: 200 mg ACH-0141625 | Segment 1: 400 mg ACH-0141625 | Segment 1: 800 mg ACH-0141625 | Segment 1: Placebo | Segment 2: 200 mg ACH-0141625 | Segment 2: 400 mg ACH-0141625 | Segment 2: 800 mg ACH-0141625
Number analyzed (Participants) | 16 | 16 | 17 | 15 | 12 | 13 | 14
percentage of participants | 75.0 | 75.0 | 64.7 | 53.3 | 100.0 | 92.3 | 100.0

8. Secondary Outcome: Segment 1 And Segment 2: Sustained Virologic Response 12 Weeks (3 Months Post-dosing) (SVR12)
Description: The percentage of virology population participants who achieved sustained virologic response (SVR), defined as HCV RNA less than the LOQ, at 12 weeks (3 months) post-dosing.
Time Frame: 3 months post-dosing
Population: Segment 2 analyzed the PPP (all randomized participants completing 12 weeks of ACH-0141625 + an extra 12 weeks of Peg/RBV) who returned for SVR12.
Measure: Number; unit: percentage of participants
Groups:
- Segment 1: 400 mg ACH-0141625: 400 mg ACH-0141625 for 28 days plus Peg-IFN alpha-2a plus RBV
  ACH-0141625: 400 mg oral capsule once daily
  Peg-IFN alpha-2a: 180 ug once a week by subcutaneous injection
  RBV: 400 mg or 600 mg (AM) and 600 mg (PM) capsules taken orally twice daily
- Segment 2: 200 mg ACH-0141625: 200 mg ACH-0141625 for 12 weeks plus Peg-IFN and RBV for up to a total of 24 or 48 weeks
  ACH-0141625: 200 mg oral capsule once daily for
  Peg-IFN alpha-2a: 180 ug once a week by subcutaneous injection
  RBV: 400 mg or 600 mg (AM) and 600 mg (PM) capsules taken orally twice daily
- Segment 2: 800 mg ACH-0141625: 800 mg ACH-0141625 for 12 weeks plus Peg-IFN and RBV for up to a total of 24 or 48 weeks
  ACH-0141625: 800 mg oral capsule once daily
  Peg-IFN Peg-IFN alpha-2a: 180 ug once a week by subcutaneous injection
  RBV: 400 mg or 600 mg (AM) and 600 mg (PM) capsules taken orally twice daily
Arm/Group | Segment 1: 200 mg ACH-0141625 | Segment 1: 400 mg ACH-0141625 | Segment 1: 800 mg ACH-0141625 | Segment 1: Placebo | Segment 2: 200 mg ACH-0141625 | Segment 2: 400 mg ACH-0141625 | Segment 2: 800 mg ACH-0141625
Number analyzed (Participants) | 16 | 16 | 17 | 15 | 10 | 13 | 13
percentage of participants | 56.3 | 56.3 | 35.3 | 40.0 | 80.0 | 76.9 | 84.5

9. Secondary Outcome: Segment 1 And Segment 2: Sustained Virologic Response 24 Weeks (6 Months Post-dosing) (SVR24)
Description: The percentage of virology population participants who achieved SVR, defined as HCV RNA less than the LOQ, 6 months post-dosing.
Time Frame: 6 months post-dosing
Population: Segment 2 analyzed the PPP (all randomized participants completing 12 weeks of ACH-0141625 plus an extra 12 weeks of Peg/RBV) who returned for SVR24
Measure: Number; unit: percentage of participants
Groups:
- Segment 2 : 800 mg ACH-0141625: 800 mg ACH-0141625 for 12 weeks plus Peg-IFN and RBV for up to a total of 48 weeks
  ACH-0141625: 800 mg oral capsule once daily for 28 days or for 12 weeks
  Peg-IFN alpha-2a: 180 ug once a week by subcutaneous injection for 48 weeks
  RBV: 400 mg or 600 mg (AM) and 600 mg (PM) capsules taken orally twice daily for 48 weeks
Arm/Group | Segment 1: 200 mg ACH-0141625 | Segment 1: 400 mg ACH-0141625 | Segment 1: 800 mg ACH-0141625 | Segment 1: Placebo | Segment 2: 200 mg ACH-0141625 | Segment 2: 400 mg ACH-0141625 | Segment 2 : 800 mg ACH-0141625
Number analyzed (Participants) | 16 | 16 | 17 | 15 | 10 | 13 | 12
percentage of participants | 62.5 | 56.3 | 35.3 | 40.0 | 70.0 | 76.9 | 83.3

10. Secondary Outcome: Segment 1 And Segment 2: HCV RNA Change From Baseline
Description: The mean change from baseline in log10 HCV RNA level by visit for the virology population
Time Frame: Week 4
Population: Efficacy analysis was performed on the virology population, which was a subset of the ITT population and included all participants who had a baseline HCV RNA result and at least 1 post-baseline HCV RNA result.
Measure: Mean (Standard Deviation); unit: log10 HCV RNA Level
Arm/Group | Segment 1: 200 mg ACH-0141625 | Segment 1: 400 mg ACH-0141625 | Segment 1: 800 mg ACH-0141625 | Segment 1: Placebo | Segment 2: 200 mg ACH-0141625 | Segment 2: 400 mg ACH-0141625 | Segment 2: 800 mg ACH-0141625
Number analyzed (Participants) | 13 | 15 | 16 | 15 | 19 | 18 | 19
log10 HCV RNA Level | -4.94 (0.993) | -4.60 (1.462) | -4.94 (1.098) | -2.22 (1.447) | -4.74 (1.072) | -5.04 (0.738) | -4.51 (0.941)

11. Secondary Outcome: Segment 1 And Segment 2: HCV RNA Change From Baseline
Description: Change from baseline in log10 HCV RNA level by visit.
Time Frame: Week 12
Population: Efficacy analysis was performed on the virology population, a subset of the ITT population, and included all participants who had a baseline HCV RNA result and at least 1 post-baseline HCV RNA result.
Measure: Mean (Standard Deviation); unit: log10 HCV RNA level
Arm/Group | Segment 1: 200 mg ACH-0141625 | Segment 1: 400 mg ACH-0141625 | Segment 1: 800 mg ACH-0141625 | Segment 1: Placebo | Segment 2: 200 mg ACH-0141625 | Segment 2: 400 mg ACH-0141625 | Segment 2: 800 mg ACH-0141625
Number analyzed (Participants) | 13 | 14 | 11 | 15 | 18 | 16 | 18
log10 HCV RNA level | -5.13 (0.518) | -4.51 (1.467) | -4.67 (1.555) | -3.48 (1.753) | -4.90 (1.104) | -5.08 (0.770) | -4.58 (0.946)

ADVERSE EVENTS:
Time Frame: Adverse event data collected through end of treatment plus 4 weeks.
Description: Treatment-emergent AEs presented: Day 1 through end of ACH-0141625/placebo treatment period plus 14 days. All serious adverse events (SAEs) reported during the study period are presented.
Groups:
- Segment 1: 200 mg ACH-0141625: 200 mg ACH-0141625 for 28 days plus Peg-IFN alpha-2a and RBV for 48 weeks
  ACH-0141625: 200 mg oral capsule
  Peg-IFN alpha-2a: 180 ug once a week by subcutaneous injection
  RBV: 400 mg or 600 mg (AM) and 600 mg (PM) capsules taken orally twice daily
- Segment 1: 400 mg ACH-0141625: 400 mg ACH-0141625 for 28 days plus Peg-IFN alpha-2a plus RBV for 48 weeks
  ACH-0141625: 400 mg oral capsule once daily
  Peg-IFN Peg-IFN alpha-2a: 180 ug once a week by subcutaneous injection
  RBV: 400 mg or 600 mg (AM) and 600 mg (PM) capsules taken orally twice daily for 48 weeks
Arm/Group | Segment 1: 200 mg ACH-0141625 | Segment 1: 400 mg ACH-0141625 | Segment 1: 800 mg ACH-0141625 | Segment 2: 200 mg ACH-0141625 | Segment 2: 400 mg ACH-0141625 | Segment 2: 800 mg ACH-0141625 | Segment 1: Placebo
Serious Adverse Events (participants affected / at risk) | 2/16 | 1/16 | 5/17 | 0/19 | 2/20 | 0/19 | 0/15
Other Adverse Events (participants affected / at risk) | 16/16 | 15/16 | 17/17 | 18/19 | 17/20 | 19/19 | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Segment 1: 200 mg ACH-0141625 (N=16) | Segment 1: 400 mg ACH-0141625 (N=16) | Segment 1: 800 mg ACH-0141625 (N=17) | Segment 2: 200 mg ACH-0141625 (N=19) | Segment 2: 400 mg ACH-0141625 (N=20) | Segment 2: 800 mg ACH-0141625 (N=19) | Segment 1: Placebo (N=15)
Ischemic Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteremia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mania (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Severe Coronary Atherosclerosis MI (death) (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Exacerbation of schizophrenia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left Lower Extremity Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Segment 1: 200 mg ACH-0141625 (N=16) | Segment 1: 400 mg ACH-0141625 (N=16) | Segment 1: 800 mg ACH-0141625 (N=17) | Segment 2: 200 mg ACH-0141625 (N=19) | Segment 2: 400 mg ACH-0141625 (N=20) | Segment 2: 800 mg ACH-0141625 (N=19) | Segment 1: Placebo (N=15)
Anaemia (Blood and lymphatic system disorders) | 0 | 4 | 3 | 2 | 1 | 2 | 3
Haemoglobinaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 2 | 3 | 2 | 5 | 5 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thyroid disorder (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abnormal sensation in eye (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 2 | 1 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 2 | 1 | 0 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2 | 1 | 2 | 1 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0 | 1 | 0
Breath odour (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 1 | 1 | 2
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 3 | 4 | 1 | 2 | 0 | 2
Dry mouth (Gastrointestinal disorders) | 2 | 2 | 0 | 0 | 1 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 1 | 1 | 3 | 1 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gingivitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lip ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 5 | 5 | 8 | 5 | 9 | 12 | 4
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2 | 2 | 2 | 2 | 1 | 1
Application site erythema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 1 | 0 | 2 | 0
Chills (General disorders) | 2 | 2 | 3 | 1 | 1 | 0 | 2
Fatigue (General disorders) | 5 | 7 | 7 | 9 | 9 | 10 | 5
Influenza like illness (General disorders) | 6 | 2 | 5 | 4 | 4 | 3 | 1
Injection site erythema (General disorders) | 2 | 2 | 4 | 1 | 0 | 0 | 3
Injection site haematoma (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Injection site irritation (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection site reaction (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Irritability (General disorders) | 3 | 3 | 2 | 2 | 2 | 5 | 1
Pain (General disorders) | 3 | 3 | 4 | 2 | 3 | 3 | 1
Pyrexia (General disorders) | 4 | 3 | 0 | 2 | 2 | 4 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 1 | 0 | 1 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Impetigo (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 0 | 0
Animal scratch (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 — Grade 3 ALT elevation occurred about Week 10. ACH-0141625 was held for 4 days, during which ALT decreased. Participant was re-challenged with ACH-0141625 for the remaining week of therapy; ALT levels continued to improve, normalizing by Week 16.
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Creatinine renal clearance decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3 | 2 | 5 | 5 | 4 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Insulin resistance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 0 | 2 | 3 | 2 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 3 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 1 | 1 | 4 | 4 | 2 | 2
Neck mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 2 | 1 | 2 | 1 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 2 | 2 | 0 | 0 | 2 | 0
Dizziness postural (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 3 | 2 | 0 | 0 | 0 | 2 | 1
Headache (Nervous system disorders) | 8 | 7 | 5 | 4 | 6 | 9 | 5
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mental impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Poor quality sleep (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Affect lability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 3 | 1 | 4 | 1 | 1
Alcohol abuse (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 0 | 2 | 2 | 0
Delusion (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 1 | 0 | 2 | 0 | 2 | 0
Depression (Psychiatric disorders) | 2 | 2 | 2 | 0 | 1 | 2 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 4 | 1 | 2 | 3 | 5 | 5 | 3
Libido decreased (Psychiatric disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0
Mania (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mood swings (Psychiatric disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0
Nervousness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sleep terror (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tearfulness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal failure chronic (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 2 | 3 | 2 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 2 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 3 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 4 | 3 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 1 | 1 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 2 | 2 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 2 | 1 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 2 | 1 | 3 | 2
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin chapped (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to submitting/presenting a manuscript or materials relating to a Study to a publisher, reviewer, or outside person, the Institution shall provide to Sponsor a copy of all such manuscripts or materials, and Sponsor shall have sixty (60) days to review and comment. The Institution shall, upon Sponsor's request, further delay publication or presentation for a period of up to one hundred twenty (120) days to allow Sponsor to protect its interests in any Sponsor Inventions.